CLINICAL TRIAL: NCT03986073
Title: A Phase IIA , Multi-center, Randomized, Double-blind, Placebo and Positive Drug Parallel Control Study of TQ-F3083 Capsules With Different Doses in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study of TQ-F3083 Capsules in Subjects With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ-F3083-II-01
Record Dates: First submitted 2019-06-09; First posted 2019-06-14 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose group (Experimental): Subjects in the low dose group administrated one TQ-F3083 capsule 10mg, one TQ-F3083 blank analog capsule and one Linagliptin blank analog tablet orally, once daily for 12 weeks.
  Interventions: Drug: TQ-F3083 capsule 10 mg; Drug: TQ-F3083 blank analog capsule; Drug: Linagliptin blank analog tablet
- High dose group (Experimental): Subjects in the high dose group administrated twoTQ-F3083 capsules 20mg and one Linagliptin blank analog tablet orally, once daily for 12 weeks.
  Interventions: Drug: TQ-F3083 capsule 20 mg; Drug: Linagliptin blank analog tablet
- Positive drug control group (Active Comparator): Subjects in the positive drug control group administrated two TQ-F3083 blank analog capsules and one Linagliptin tablet orally, once daily for 12 weeks.
  Interventions: Drug: TQ-F3083 blank analog capsule; Drug: Linagliptin tablet
- Placebo group (Placebo Comparator): Subjects in the placebo group administrated two TQ-F3083 blank analog capsules and one Linagliptin blank analog tablet orally, once daily for 12 weeks.
  Interventions: Drug: TQ-F3083 blank analog capsule; Drug: Linagliptin blank analog tablet

INTERVENTIONS:
Drug: TQ-F3083 capsule 10 mg — Subjects in the low dose group administrated TQ-F3083 capsule 10mg, once daily for 12 weeks.
  Arms: Low dose group
Drug: TQ-F3083 capsule 20 mg — Subjects in the high dose group administrated TQ-F3083 capsule 20 mg, once daily for 12 weeks.
  Arms: High dose group
Drug: TQ-F3083 blank analog capsule — Subjects administrated one TQ-F3083 blank analog capsule orally, once daily for 12 weeks.
  Arms: Low dose group
Drug: TQ-F3083 blank analog capsule — Subjects administrated two TQ-F3083 blank analog capsules orally, once daily for 12 weeks.
  Arms: Placebo group; Positive drug control group
Drug: Linagliptin blank analog tablet — Subjects administrated one Linagliptin blank analog tablet orally, once daily for 12 weeks.
  Arms: High dose group; Low dose group; Placebo group
Drug: Linagliptin tablet — Subjects in the positive drug control group administrated one Linagliptin tablet orally, once daily for 12 weeks.
  Arms: Positive drug control group

SUMMARY:
TQ-F3083 capsule is a new type inhibitor of DPP-IV, which is currently a very effective target for the treatment of type 2 diabetes mellitus at clinical. In addition, it can promote insulin secretion with low potential toxicity, and half-life is shorter than Linagliptin.

ELIGIBILITY:
Inclusion Criteria:

1.Understood and signed an informed consent form; 2.18 and 70 years old; 3.Body mass index (BMI) of 19 to 37.5 kg/m2; 4.Type 2 diabetes mellitus confirmed at least 6 weeks before screen by WHO (1999) diabetes mellitus diagnostic criteria; 5.Has inadequate glycemic control on diet/exercise therapy and irregular use hypoglycemic agents before screening, HbA1c ≥7.0% and ≤10.0% ; Has regular hypoglycemic agents with stable dose within 6 weeks before screening, HbA1c ≥7.0% and ≤9 %; 6.PFG ≤ 13.3 mmol / L; 7. Adequate laboratory inspection standards.

Exclusion Criteria:

1. Has any contraindications, allergies or hypersensitivity for taking research medication ;
2. Has used at lest two oral medications to treat diabetes mellitus 6 weeks before screening;
3. Has other endocrine-related history or evidence before screening;
4. Has history of organ transplantation;
5. Has mental or neurological diseases;
6. Has received systemic corticosteroids within 2 weeks;
7. Has received GLP-1 analogues, DPP-4 inhibitors or anti-obesity drugs 3 months ;
8. Has alcohol abuse history within 6 months before screening;
9. Has participated in any clinical trial within 3 months;
10. Has received blood transfusions, or blood donation ≥ 400 mL , or got severe blood loss ≥ 400 mL within 8 weeks;
11. Pregnant or lactating woman.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | up to approximately 15 weeks
  Changes in HbA1c compared with baseline after 12 weeks of treatment

SECONDARY OUTCOMES:
Fasting plasma glucose (FPG) | up to approximately 15 weeks
  Changes in FPG compared with baseline after 12 weeks of treatment
2 hours-postprandial blood sugar (2h-PPG） | up to approximately 15 weeks
  Changes in 2h-PPG compared with baseline after 12 weeks of treatment
Weight | up to approximately 7, 11, 15 weeks
  Changes in weight compared with baseline after 4, 8, 12 weeks of treatment
HbA1c | up to approximately 15 weeks
  The proportion of patients with HbA1c less than 7% after 12 weeks of treatment
HbA1c | up to approximately 15 weeks
  The proportion of patients with HbA1c reduced at least 0.5% after 12 weeks of treatment
DPP-4 activity ( dipeptidyl peptidase-4) | baseline up to 4, 8, 12 weeks
  changes in DPP-4 activity compared with baseline after 4, 8, 12 weeks of treatment
GLP-1 (glucagon-like peptide-1) | baseline up to 4, 8, 12 weeks
  changes in DPP-4 activity GLP-1 concentrations compared with baseline after 4, 8, 12 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The Second Affiliated Hospital of Chongqing Medical Uversity, Chongqing, Chongqing Municipality
  - Chongqing General Hospital, UCAS, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Yuncheng Central Hospital, Jinan, Shandong
  - Jincheng Geberal Hospital, Jincheng, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan